CLINICAL TRIAL: NCT01600937
Title: Italian Diabetes and Exercise Study 2 - A Long-term Behavioural Intervention for Adoption and Maintenance of a Physically Active Lifestyle
Brief Title: Italian Diabetes and Exercise Study 2
Acronym: IDES-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metabolic Fitness Association, Italy (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giuseppe Pugliese, MD, PhD, Metabolic Fitness Association, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MFA-12-01
Record Dates: First submitted 2012-05-16; First posted 2012-05-17 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes
Keywords: diabetes mellitus; diabetes education; behavioral therapy; behavior modification; physical activity; supervised exercise; physical fitness; HbA1c; modifiable cardiovascular risk factors; quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Standard care including physician recommendations for daily PA
- Exercise (Experimental): Theoretical & practical exercise counseling including 2 sessions/ per wk for 1 month of supervised exercise training
  Interventions: Behavioral: Theoretical & practical exercise counseling

INTERVENTIONS:
Behavioral: Theoretical & practical exercise counseling — 2 sessions/ per wk for 1 month
  Arms: Exercise

SUMMARY:
Current guidelines recommend supervised mixed (aerobic+resistance) physical activity to ensure optimal benefits to control blood glucose, lipids, blood pressure, and other cardiovascular risk and to minimize injuries. However, these guidelines are difficult to put into action for a number of barriers and poor long-term patient compliance. This project will assess the effect of a behavioral intervention strategy on the promotion and maintenance of physical activity in type 2 diabetes.

DETAILED DESCRIPTION:
An increasing prevalence of type 2 diabetes is associated with an aging population, a significant rise in the prevalence of obesity, and a sedentary lifestyle. In Italy, prevalence of diabetes is approximately 6%, with 90-95% of diabetic subjects having type 2. Strong evidence supports the importance of physical activity in the management of type 2 diabetes. However, current guidelines are difficult to put into action in this target population because of barriers and poor patient long-term compliance so it is difficult even identify the best strategies for physical activity behavior change. Existing studies employ small groups and clinically-based approaches with limited theoretical grounding for recommended health behavior change. Most fail to offer practical, sustainable, economically viable solutions, with documented long-term intervention efficacy. This study proposes to monitor any objective measurable changes in LTPA over a 3-year period after behavioral interventions (Physician recommendations for daily PA with and without supervised exercise training including individual theoretic & practical counseling). Hopefully, such behavioral intervention would offer a feasible procedure for long-term maintenance of physical activity and thus meet the call for a change of paradigm to move beyond the limited clinical focus by including theoretically population-based and "real-life" approaches for the management Type 2 Diabetes.

After the selection for eligibility and a run-in period, patients will be randomized in two groups: 1) exercise (EXE) group receiving theoretical & practical exercise counseling including 2 sessions/ per wk for 1 month of supervised exercise training; and 2) control (CON) group receiving standard care including general physician recommendations for daily PA. Changes in physical activity behavior will be quantified using an accelerometer, in addition to a daily diary.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. Age 40 to 80 years at screening
3. BMI >27<40 kg/m2
4. Sedentary for at least 6 months
5. Treated with prescribed diet and/or OHA and insulin
6. Able to walk for 1.6 Km unaided.
7. Eligible after positive outcome of cardiac evaluation

Exclusion Criteria:

1. All patients with a history of central nervous dysfunction such as hemiparesis, myelopathies, cerebral ataxia, significant musculoskeletal deformities such as an amputation, dysmetria or scoliosis, patients with movement abnormalities or arthritis limited by pain when exercising
2. A history of clinical evidence of severe cardiovascular disease which may limit or be a contraindication for exercise
3. Clinical evidence of vestibular dysfunction
4. Angina and related symptoms
5. Postural hypotension defined as a fall in arterial blood pressure when changing position of >20 mmHg (systole) or >10 mmHg (diastole
6. History of plantar sores

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-10; Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Physical Activity Behavior | 3 years
  Volume of physical activity in METs-hr/wk; sedentary time; time spent in moderate-to-vigorous physical activity

SECONDARY OUTCOMES:
Physical fitness | 3 years
  Physical fitness (Cardiorespiratory, fitness, muscle strength, hip and trunk flexibility)
Modifiable cardiovascular risk factors | 3 years
  Modifiable cardiovascular risk factors (HbA1c, lipids, blood pressure, C-reactive protein, CHD 10-year risk scores)
Health related quality of life | 3 years
  Quality of life (Physical and mental SF-36 scores)
Musculo-skeletal disturbances | 3 years
  Musculo-skeletal symproms and scores

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Balducci, MD, Study Director — Sant'Andrea Hospital, Diabetes Unit
Locations (1):
- University of Rome La Sapienza, Department of Clinical and Molecular Medicine, Sant'Andrea Hospital, Diabetes Unit, Rome, RM, Italy

REFERENCES:
- [Background] Balducci S, Zanuso S, Cardelli P, Salvi L, Mazzitelli G, Bazuro A, Iacobini C, Nicolucci A, Pugliese G; Italian Diabetes Exercise Study (IDES) Investigators. Changes in physical fitness predict improvements in modifiable cardiovascular risk factors independently of body weight loss in subjects with type 2 diabetes participating in the Italian Diabetes and Exercise Study (IDES). Diabetes Care. 2012 Jun;35(6):1347-54. doi: 10.2337/dc11-1859. Epub 2012 Mar 7. PMID 22399699
- [Background] Nicolucci A, Balducci S, Cardelli P, Cavallo S, Fallucca S, Bazuro A, Simonelli P, Iacobini C, Zanuso S, Pugliese G; Italian Diabetes Exercise Study Investigators. Relationship of exercise volume to improvements of quality of life with supervised exercise training in patients with type 2 diabetes in a randomised controlled trial: the Italian Diabetes and Exercise Study (IDES). Diabetologia. 2012 Mar;55(3):579-88. doi: 10.1007/s00125-011-2425-9. Epub 2012 Jan 11. PMID 22234648
- [Background] Balducci S, Zanuso S, Pugliese G, Church T, Sigal RJ. Diet or diet plus physical activity in patients with early type 2 diabetes. Lancet. 2011 Dec 17;378(9809):2066; author reply 2067-8. doi: 10.1016/S0140-6736(11)61891-6. No abstract available. PMID 22177504
- [Background] Nicolucci A, Balducci S, Cardelli P, Zanuso S, Pugliese G; Italian Diabetes Exercise Study (IDES) Investigators. Improvement of quality of life with supervised exercise training in subjects with type 2 diabetes mellitus. Arch Intern Med. 2011 Nov 28;171(21):1951-3. doi: 10.1001/archinternmed.2011.561. No abstract available. PMID 22123809
- [Background] Balducci S, Zanuso S, Cardelli P, Salerno G, Fallucca S, Nicolucci A, Pugliese G; Italian Diabetes Exercise Study (IDES) Investigators. Supervised exercise training counterbalances the adverse effects of insulin therapy in overweight/obese subjects with type 2 diabetes. Diabetes Care. 2012 Jan;35(1):39-41. doi: 10.2337/dc11-1450. Epub 2011 Oct 19. PMID 22011409
- [Background] Balducci S, Zanuso S, Nicolucci A, De Feo P, Cavallo S, Cardelli P, Fallucca S, Alessi E, Fallucca F, Pugliese G; Italian Diabetes Exercise Study (IDES) Investigators. Effect of an intensive exercise intervention strategy on modifiable cardiovascular risk factors in subjects with type 2 diabetes mellitus: a randomized controlled trial: the Italian Diabetes and Exercise Study (IDES). Arch Intern Med. 2010 Nov 8;170(20):1794-803. doi: 10.1001/archinternmed.2010.380. PMID 21059972
- [Background] Balducci S, Zanuso S, Nicolucci A, Fernando F, Cavallo S, Cardelli P, Fallucca S, Alessi E, Letizia C, Jimenez A, Fallucca F, Pugliese G. Anti-inflammatory effect of exercise training in subjects with type 2 diabetes and the metabolic syndrome is dependent on exercise modalities and independent of weight loss. Nutr Metab Cardiovasc Dis. 2010 Oct;20(8):608-17. doi: 10.1016/j.numecd.2009.04.015. Epub 2009 Aug 19. PMID 19695853
- [Background] Pugliese G, Zanuso S, Alessi E, Simonelli P, Fallucca S, Fallucca F, Balducci S. Self glucose monitoring and physical exercise in diabetes. Diabetes Metab Res Rev. 2009 Sep;25 Suppl 1:S11-7. doi: 10.1002/dmrr.982. PMID 19662620
- [Background] Balducci S, Zanuso S, Fernando F, Fallucca S, Fallucca F, Pugliese G; Italian Diabetes Exercise Study (IDES) Group. Physical activity/exercise training in type 2 diabetes. The role of the Italian Diabetes and Exercise Study. Diabetes Metab Res Rev. 2009 Sep;25 Suppl 1:S29-33. doi: 10.1002/dmrr.985. PMID 19662617
- [Background] Zanuso S, Balducci S, Gutierrez AJ, Bergamin M, Pugliese G. Similar energy expenditure from resistance training at moderate and vigorous intensity in subjects with type 2 diabetes. Diabetes Res Clin Pract. 2009 Sep;85(3):e40-1. doi: 10.1016/j.diabres.2009.05.003. Epub 2009 Jun 4. No abstract available. PMID 19500870
- [Background] Zanuso S, Jimenez A, Pugliese G, Corigliano G, Balducci S. Exercise for the management of type 2 diabetes: a review of the evidence. Acta Diabetol. 2010 Mar;47(1):15-22. doi: 10.1007/s00592-009-0126-3. Epub 2009 Jun 3. PMID 19495557
- [Background] Balducci S, Zanuso S, Massarini M, Corigliano G, Nicolucci A, Missori S, Cavallo S, Cardelli P, Alessi E, Pugliese G, Fallucca F; Italian Diabetes Exercise Study (IDES) Group. The Italian Diabetes and Exercise Study (IDES): design and methods for a prospective Italian multicentre trial of intensive lifestyle intervention in people with type 2 diabetes and the metabolic syndrome. Nutr Metab Cardiovasc Dis. 2008 Nov;18(9):585-95. doi: 10.1016/j.numecd.2007.07.006. Epub 2007 Dec 3. PMID 18061415
- [Background] Balducci S, Alessi E, Cardelli P, Cavallo S, Fallucca F, Pugliese G. Effects of different modes of exercise training on glucose control and risk factors for complications in type 2 diabetic patients: a meta-analysis: response to Snowling and Hopkins. Diabetes Care. 2007 Apr;30(4):e25; author reply e26. doi: 10.2337/dc06-2495. No abstract available. PMID 17392536
- [Derived] Balducci S, Haxhi J, Vitale M, Mattia L, Calvi F, Marini M, Ciocca E, Auccello F, Gentile A, Sacchetti M, Orlando G, Zanuso S, Nicolucci A, Pugliese G; Italian Diabetes and Exercise Study 2 (IDES_2) Investigators. Effect of a behavioral counseling for adoption and maintenance of a physically active lifestyle on long-term mortality in people with type 2 diabetes: post hoc analysis of the Italian Diabetes and Exercise Study_2. Nat Commun. 2026 Jan 22. doi: 10.1038/s41467-026-68618-7. Online ahead of print. PMID 41571659
- [Derived] Balducci S, Haxhi J, Vitale M, Mattia L, Sacchetti M, Orlando G, Cardelli P, Iacobini C, Bollanti L, Conti F, Zanuso S, Nicolucci A, Pugliese G; Italian Diabetes and Exercise Study 2 (IDES_2) Investigators. Sustained increase in physical fitness independently predicts improvements in cardiometabolic risk profile in type 2 diabetes. Diabetes Metab Res Rev. 2023 Sep;39(6):e3671. doi: 10.1002/dmrr.3671. Epub 2023 Jun 14. PMID 37312666
- [Derived] Balducci S, Haxhi J, Sacchetti M, Orlando G, Cardelli P, Vitale M, Mattia L, Iacobini C, Bollanti L, Conti F, Zanuso S, Nicolucci A, Pugliese G; Italian Diabetes and Exercise Study 2 (IDES_2) Investigators. Relationships of Changes in Physical Activity and Sedentary Behavior With Changes in Physical Fitness and Cardiometabolic Risk Profile in Individuals With Type 2 Diabetes: The Italian Diabetes and Exercise Study 2 (IDES_2). Diabetes Care. 2022 Jan 1;45(1):213-221. doi: 10.2337/dc21-1505. PMID 34728529
- [Derived] Nicolucci A, Haxhi J, D'Errico V, Sacchetti M, Orlando G, Cardelli P, Vitale M, Bollanti L, Conti F, Zanuso S, Lucisano G, Balducci S, Pugliese G; Italian Diabetes and Exercise Study 2 (IDES_2) Investigators. Effect of a Behavioural Intervention for Adoption and Maintenance of a Physically Active Lifestyle on Psychological Well-Being and Quality of Life in Patients with Type 2 Diabetes: The IDES_2 Randomized Clinical Trial. Sports Med. 2022 Mar;52(3):643-654. doi: 10.1007/s40279-021-01556-0. Epub 2021 Oct 1. PMID 34599476
- [Derived] Balducci S, D'Errico V, Haxhi J, Sacchetti M, Orlando G, Cardelli P, Vitale M, Bollanti L, Conti F, Zanuso S, Lucisano G, Nicolucci A, Pugliese G; Italian Diabetes and Exercise Study 2 (IDES_2) Investigators. Effect of a Behavioral Intervention Strategy on Sustained Change in Physical Activity and Sedentary Behavior in Patients With Type 2 Diabetes: The IDES_2 Randomized Clinical Trial. JAMA. 2019 Mar 5;321(9):880-890. doi: 10.1001/jama.2019.0922. PMID 30835309
- [Derived] Balducci S, D'Errico V, Haxhi J, Sacchetti M, Orlando G, Cardelli P, Vitale M, Bollanti L, Conti F, Zanuso S, Nicolucci A, Pugliese G; Italian Diabetes and Exercise Study 2 (IDES-_2) Investigators. Effect of a Behavioral Intervention Strategy for Adoption and Maintenance of a Physically Active Lifestyle: The Italian Diabetes and Exercise Study 2 (IDES_2): A Randomized Controlled Trial. Diabetes Care. 2017 Nov;40(11):1444-1452. doi: 10.2337/dc17-0594. Epub 2017 Aug 18. PMID 28821576
- [Derived] Balducci S, D'Errico V, Haxhi J, Sacchetti M, Orlando G, Cardelli P, Di Biase N, Bollanti L, Conti F, Zanuso S, Nicolucci A, Pugliese G; Italian Diabetes and Exercise Study 2 (IDES_2) Investigators. Level and correlates of physical activity and sedentary behavior in patients with type 2 diabetes: A cross-sectional analysis of the Italian Diabetes and Exercise Study_2. PLoS One. 2017 Mar 14;12(3):e0173337. doi: 10.1371/journal.pone.0173337. eCollection 2017. PMID 28291838
- [Derived] Balducci S, Sacchetti M, Haxhi J, Orlando G, Zanuso S, Cardelli P, Cavallo S, D'Errico V, Ribaudo MC, Di Biase N, Salvi L, Vitale M, Bollanti L, Conti FG, Nicolucci A, Pugliese G; Italian Diabetes and Exercise Study 2 (IDES_2) Investigators. The Italian Diabetes and Exercise Study 2 (IDES-2): a long-term behavioral intervention for adoption and maintenance of a physically active lifestyle. Trials. 2015 Dec 11;16:569. doi: 10.1186/s13063-015-1088-0. PMID 26651484
- See also: Study protocol — http://www.metabolicfitness.it/